CLINICAL TRIAL: NCT01544101
Title: A Nutritional Intervention for Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WCCR-ARTH1
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Diet, Vegetarian; Diet, Fat-Restricted; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegan Diet (Experimental)
  Interventions: Other: Vegan Diet
- Supplement (Placebo Comparator)
  Interventions: Dietary Supplement: dietary supplement omega3 fatty acids aand vitamins

INTERVENTIONS:
Other: Vegan Diet — Vegan diet, which is devoid of animal products and minimal in fat
  Arms: Vegan Diet
Dietary Supplement: dietary supplement omega3 fatty acids aand vitamins — mixture of omega3 fatty acids aand vitamins
  Arms: Supplement

SUMMARY:
The purpose of the study is to assess whether, in individuals with rheumatoid arthritis, a low-fat, vegan diet improves pain and other subjective symptoms more effectively than a control supplement or a placebo. The principal measure is pain as measured by Visual Analog Scale (VAS) and disease activity as measured by number of painful swollen and tender joints, respectively. The study duration is 36 weeks.

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian diets and certain nutritional supplements can help reduce pain and also reduce the need for pain medications for some people. The investigators will ask about 100 people to participate. All of them will get a low-fat, vegan diet and a nutritional supplement (mixture of omega-3 oils and vitamin E or a placebo), although some will get the diet first, and others will get the supplement first. This order in which they will get the diet and the supplement will be determined randomly, that is, by chance (like the toss of a coin). The principal measure is pain as measured by Visual Analog Scale (VAS) and disease activity as measured by number of painful swollen and tender joints, respectively. The study duration is 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of rheumatoid arthritis, as defined below.

   A diagnosis of rheumatoid arthritis is based on 2010 ACR / EULAR Rheumatoid Arthritis Classification Criteria. Classification as "definite RA" is based on the confirmed presence of synovitis in at least 1 joint, absence of an alternative diagnosis that better explains the synovitis, and achievement of a total score of 6 or greater (of a possible 10): 24

   Joint involvement, designating the metacarpophalangeal joints, proximal interphalangeal joints, the interphalangeal joint of the thumb, second through third metatarsophalangeal joint and wrist as small joints, and elbows, hip joints and knees as large joints:
   * Involvement of 1 large joint gives 0 points
   * Involvement of 2-10 large joints gives 1 point
   * Involvement of 1-3 small joints (with or without involvement of large joints) gives 2 points
   * Involvement of4-10 small joints (with or without involvement of large joints) gives 3 points
   * Involvement of more than 10 joints (with involvement of at least 1 small joint) gives 5 points

   Serological parameters - including the rheumatoid factor as well as anti-citrullinated protein antibody (ACPA):
   * Negative RF and negative ACPA gives 0 points
   * Low-positive RF or low-positive ACPA gives 2 points
   * High-positive RF or high-positive ACPA gives 3 points Acute phase reactants: 1 point for elevated erythrocyte sedimentation rate (ESR) or elevated C-reactive protein (CRP) value Duration of arthritis: 1 point for symptoms lasting six weeks or longer
2. Continuing or recurring pain (i.e., joint pain daily, unless on pain medication).
3. Age at least 18 years
4. Ability and willingness to participate in all components of the study
5. Willingness to be assigned to either the diet group or supplement group
6. Pain medications unchanged within last 6 weeks.

Exclusion Criteria:

1. < 18 years of age
2. Rheumatoid arthritis for more than 6 years
3. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
4. Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
5. Pregnancy
6. Unstable medical or psychiatric illness
7. Likely to be disruptive in group sessions (as determined by research staff)
8. Already following a low-fat, vegan diet
9. Lack of English fluency
10. Inability to maintain current medication regimen
11. Inability or unwillingness to participate in all components of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pain Score | Baseline and 4 months
  will be measured by visual analog scale
Disease Activity score | Baseline and 4 months
  measured by number of painful, swollen and tender joints

SECONDARY OUTCOMES:
Quality of Life | Baseline and 4 months
  measured by a modified health assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Barnard ND, Levin S, Crosby L, Flores R, Holubkov R, Kahleova H. A Randomized, Crossover Trial of a Nutritional Intervention for Rheumatoid Arthritis. Am J Lifestyle Med. 2022 Apr 3;19(2):266-275. doi: 10.1177/15598276221081819. eCollection 2025 Feb. PMID 39981557